CLINICAL TRIAL: NCT01851018
Title: Match Pair Analysis Study, Comparing Toxicities Between 2 Treatment Regiments Including Neo-adjuvant Hormonal Therapy Plus Hypofractionated RT With HDR Brachytherapy Boost Compare to Our Current Clinical Standard Approach at CHU de Quebec
Brief Title: Toxicity Comparison Between Hypofractionated Radiotherapy With HDR Brachytherapy Boost Versus Standard Treatment
Acronym: HyBraFi
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, André-Guy Martin, André-Guy Martin MD MSC FRCP(C) Radio-oncologue, Curiethérapeute Professeur Associé, Université Laval, L'Hôtel-Dieu de Québec du CHUQ, CHU de Quebec-Universite Laval
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H12-03-90; HYBRAFI (Other: CHUdeQuebec)
Record Dates: First submitted 2012-11-27; First posted 2013-05-10 (Estimated); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; brachytherapy; hypofractionated radiation therapy; hormonal therapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Radiation (hypo fractionation)
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypofraction (Experimental): Patient reported toxicities related to Hypofraction radiation treatment (3 Gy daily, 5 fractions per week) up to a total of 36 Gy to the prostate (+/- seminal vesicles) plus brachytherapy boost (15 Gy in a single fraction) with 4 months neo-adjuvant firmagon (240 mg given as two subcutaneous injections of 120 mg at a concentration of 40 mg/mL as a starting dose with a maintenance dose of 80 mg given as one subcutaneous injection at a concentration of 20 mg/mL administered every 28 days).
  Interventions: Radiation: Hypofraction
- Standard (Active Comparator): Patient reported toxicities related to the Standard radiation treatment (2 Gy daily, 5 fractions per week) up to a total of 44 Gy to the prostate (+/- seminal vesicles) plus brachytherapy boost (15 Gy in a single fraction) with 4 months neo-adjuvant LHRH agonists.
  Interventions: Radiation: Standard

INTERVENTIONS:
Radiation: Hypofraction — Patient reported toxicities related to Hypofraction radiation treatment (3 Gy daily, 5 fractions per week) up to a total of 36 Gy to the prostate (+/- seminal vesicles) plus brachytherapy boost (15 Gy in a single fraction) with 4 months neo-adjuvant firmagon (240 mg given as two subcutaneous injections of 120 mg at a concentration of 40 mg/mL as a starting dose with a maintenance dose of 80 mg given as one subcutaneous injection at a concentration of 20 mg/mL administered every 28 days).
  Arms: Hypofraction
Radiation: Standard — Patient reported toxicities related to the Standard radiation treatment (2 Gy daily, 5 fractions per week) up to a total of 44 Gy to the prostate (+/- seminal vesicles) plus brachytherapy boost (15 Gy in a single fraction) with 4 months neo-adjuvant LHRH agonists
  Arms: Standard

SUMMARY:
The purpose of this study is to compare toxicities between 2 external beam radiation fractionation schemes plus a brachytherapy boost for prostate cancer. Our current standard use a 2 Gy per fraction schedule which is compare to the experimental hypofractionated 3 Gy per day approach with neo adjuvant hormonal therapy. It will demonstrate the feasibility and safety of such a treatment regimen in prostate cancer. It may also set base for a larger randomized trial.

DETAILED DESCRIPTION:
30 patients with intermediate / extensive low risk (all core biopsies involvements > 50%) prostate cancer (not necessitating to treat the nodal regions) will be included in this study. Patient stage T1 - T2, Gleason score ≤ 7, prostate-specific antigen (PSA) ≤ 20 will be considered.

Fiducial gold markers will be introduced in the prostate 1-week before the CT planning. 36 gray (Gy) in 12 fractions using intensity-modulated radiation therapy (IMRT) will be administered to the prostate (margins of 0,5cm) +/- first centimeter of the seminal vesicles.

Brachytherapy boost (15 Gy x 1) dosimetric parameters should respect our current standard (Prostate V100 > 90% and V150 ≤ 40%, V200 ≤ 15%, Urethra V125 ≤ 1 cc, Rectum V75 ≤ 1cc, Bladder V75 ≤ 1cc). Short course (4 months) hormonal therapy (Degarelix) will be administered to the patient based upon recommended litterature11, 12.

Genitourinary (GU), GI and Sexual toxicity will be self reported. QOL questionnaires will be given to the patients to be answered. Results will be monitored and compared to our currently used standard fractionation regiment.

Follow-up will be scheduled 6 weeks after the implant and every 4 months for the first year, every 6 months for the second year 2 to 5, and on a yearly basis after 5 years. PSA & testosterone tests will be done every 3 months for the first 3 years, every 6 months on years 4 and 5, and yearly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* 30 patients
* intermediate / extensive low risk (all core biopsies involvements > 50%)
* prostate cancer (not necessitating to treat the nodal regions)
* Patient stage T1 - T2,
* Gleason score ≤ 7,
* PSA ≤ 20 will be considered

Exclusion Criteria:

* patient unfit for biopsy or brachytherapy
* high or low risk prostate cancer

Ages: 18 Years to 95 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-05; Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate and compare toxicity changes through follow-up between our study population and a reference group in regards to Median international prostate symptoms scores (IPSS). | baseline, 6 weeks post-implant, and at 4,8,12 months
  Comparison of the patient reported IPSS scores through the follow-up between each treatment group.
Evaluate and compare toxicity changes through follow-up between our study population and a reference group in regards to gastro-intestinal (GI) toxicity score. | baseline, 6 weeks post-implant, and at 4,8,12 months
  Comparison of the patient reported Gastro-intestinal toxicity scores through the follow-up between each treatment group.
Evaluate and compare toxicity changes through follow-up between our study population and a reference group in regards to Sexual toxicity (EPIC or SHIM) score. | baseline, 6 weeks post-implant, and at 4,8,12 months
  Comparison of the patient reported Sexual toxicity (EPIC or SHIM) scores through the follow-up between each treatment group.

SECONDARY OUTCOMES:
Evaluate and compare biochemical disease free survival being non inferior to comparative cohort | 5 years
  biochemical disease free survival (Phoenix definition)

CONTACTS AND LOCATIONS:
Overall Officials: Andre-Guy Martin, MD MSc, Principal Investigator — CHUQ L'Hotel Dieu de Quebec
Locations (1):
- CHUdeQuebec, Québec, Canada

REFERENCES:
- [Derived] De Bari B, Daidone A, Alongi F. Is high dose rate brachytherapy reliable and effective treatment for prostate cancer patients? A review of the literature. Crit Rev Oncol Hematol. 2015 Jun;94(3):360-70. doi: 10.1016/j.critrevonc.2015.02.003. Epub 2015 Feb 17. PMID 25819287